CLINICAL TRIAL: NCT05874245
Title: PERIOPERATIVE EFFECTS OF ORAL DEXMEDETOMIDINE, KETAMINE, OR MIDAZOLAM PREMEDICATION IN CHILDREN UNDERGOING ADENOTONSILLECTOMY
Brief Title: Effect of Oral Dexmedetomidine, Ketamine, Or Midazolam as Preioperative Medications.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmed elsayed mahmoud abousayar, Principal Investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 11\2022 ANES 15
Record Dates: First submitted 2023-04-05; First posted 2023-05-24 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: The study will be a prospective randomized double-blind study. Patients will be randomized into three groups using a closed envelope technique in sequentially numbered opaque envelopes that will be opened by an anesthesiologist not involved in the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group D; oral Dexmedetomidine (Experimental): will receive 4 micrograms/kg oral Dexmedetomidine diluted in paracetamol [Paracetamol syrup 150 mg/5ml] at a dose of 15 mg/kg given 45 minutes before the induction of anaesthesia.
  Interventions: Drug: oral Dexmedetomidine
- Group K; oral ketamine group (Experimental): will receive 6 mg/kg oral Ketamine diluted in paracetamol [Paracetamol syrup 150 mg/5ml] at a dose of 15 mg/kg 45 minutes before the induction of anaesthesia.
  Interventions: Drug: oral ketamine
- Group M; oral Midazolam group (Experimental): will receive 0.3 mg/kg (maximum 20 mg) oral Midazolam diluted in paracetamol [Paracetamol syrup 150 mg/5ml] at a dose of 15 mg/kg given 45 minutes before the induction of anaesthesia.
  Interventions: Drug: oral Midazolam

INTERVENTIONS:
Drug: oral Dexmedetomidine — will receive 4 micrograms/kg oral Dexmedetomidine diluted in paracetamol [Paracetamol syrup 150 mg/5ml] at a dose of 15 mg/kg given 45 minutes before the induction of anaesthesia
  Arms: Group D; oral Dexmedetomidine
Drug: oral ketamine — will receive 6 mg/kg oral ketamine diluted in paracetamol [Paracetamol syrup 150 mg/5ml] at a dose of 15 mg/kg 45 minutes before the induction of anaesthesia
  Arms: Group K; oral ketamine group
Drug: oral Midazolam — will receive 0.3 mg/kg (maximum 20 mg) oral Midazolam diluted in paracetamol [Paracetamol syrup 150 mg/5ml] at a dose of 15 mg/kg given 45 minutes before the induction of anaesthesia
  Arms: Group M; oral Midazolam group

SUMMARY:
Anxiety preceding surgery results in hemodynamic instability, metabolic side effects, increased post-operative pain, and agitation during emergence. Therefore, pharmacological interventions are used to reduce pre-operative anxiety and enhance anesthetic induction without delaying recovery. The premedication must be administered in a manner that is safe, painless, and without significant adverse effects.

In children, the incidence of emergency agitation or delirium after general anesthesia ranges from 10% to 80% and significantly increases the incidence of other complications after anesthesia, such as self-injury, prolonged postanesthesia care unit (PACU) stay, frustration of parents and care providers.

Numerous pharmacological and non-pharmacological techniques, including sedative premedication, parental presence, and training programs for participants and their parents, have been investigated to reduce anxiety and enhance compliance during anesthesia induction.

An ideal premedication prescription should sedate a child to facilitate separation from parents, thus simplifying anesthesia induction and creating a pleasant surgical experience for both children and parents. [5]

Anxiolysis is the major objective of premedication in children, as it facilitates separation from parents and facilitates the induction of anesthesia.

Premedication may also induce amnesia, the prevention of physiologic stress, vagolysis, a decrease in total anesthetic requirements, a lower likelihood of aspiration, decreased salivation and secretions, antiemesis, and analgesia. All drugs have the potential to make people sleepy and slow their breathing, so they must be given with extreme care and closely watched.

Ketamine is a useful sedative and analgesic for preventing preoperative anxiety in children; it exerts its analgesic effect through the reversible antagonist action of N-methyl-D-aspartate receptors. It has analgesic and sedative effects in different doses of administration. Ketamine is often administered orally and is αreported to be safe and effective in pediatric patients.

An effective sedative and analgesic with minimal respiratory depressive effects is dexmedetomidine, an α2-adrenoceptor agonist. It also reduces the hemodynamic stress response due to its sympatholytic effect. These characteristics make it a possible anesthetic premedication.

Midazolam, a water-soluble benzodiazepine, is commonly used as a preanesthetic medicine in children due to its several favorable effects: sedation, anxiolysis, antegrade amnesia, rapid onset, and brief duration of action.

Adenoidectomy and/or tonsillectomy are the most common surgical procedures done on children.

Hence, the present study will be conducted to objectively evaluate, the perioperative effects of oral dexmedetomidine, ketamine, or midazolam premedication in patients undergoing adenotonsillectomy.

DETAILED DESCRIPTION:
Anxiety preceding surgery results in hemodynamic instability, metabolic side effects, increased post-operative pain, and agitation during emergence. Therefore, pharmacological interventions are used to reduce pre-operative anxiety and enhance anesthetic induction without delaying recovery. The premedication must be administered in a manner that is safe, painless, and without significant adverse effects.

In children, the incidence of emergency agitation or delirium after general anesthesia ranges from 10% to 80% and significantly increases the incidence of other complications after anesthesia, such as self-injury, prolonged postanesthesia care unit (PACU) stay, frustration of parents and care providers.

Numerous pharmacological and non-pharmacological techniques, including sedative premedication, parental presence, and training programs for participants and their parents, have been investigated to reduce anxiety and enhance compliance during anesthesia induction.

An ideal premedication prescription should sedate a child to facilitate separation from parents, thus simplifying anesthesia induction and creating a pleasant surgical experience for both children and parents.

Anxiolysis is the major objective of premedication in children, as it facilitates separation from parents and facilitates the induction of anesthesia.

Premedication may also induce amnesia, the prevention of physiologic stress, vagolysis, a decrease in total anesthetic requirements, a lower likelihood of aspiration, decreased salivation and secretions, anti-emesis, and analgesia. All drugs have the potential to make people sleepy and slow their breathing, so they must be given with extreme care and closely watched.

Ketamine is a useful sedative and analgesic for preventing preoperative anxiety in children; it exerts its analgesic effect through the reversible antagonist action of N-methyl-D-aspartate receptors. It has analgesic and sedative effects in different doses of administration. Ketamine is often administered orally and is αreported to be safe and effective in pediatric patients.

An effective sedative and analgesic with minimal respiratory depressive effects is dexmedetomidine, an α2-adrenoceptor agonist. It also reduces the hemodynamic stress response due to its sympatholytic effect. These characteristics make it a possible anesthetic premedication. Midazolam, a water-soluble benzodiazepine, is commonly used as a preanesthetic medicine in children due to its several favorable effects: sedation, anxiolysis, antegrade amnesia, rapid onset, and brief duration of action.

Adenoidectomy and/or tonsillectomy are the most common surgical procedures done on children.

Hence, the present study will be conducted to objectively evaluate, the perioperative effects of oral dexmedetomidine, ketamine, or midazolam premedication in patients undergoing adenotonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

* All patients within the age range of 3 to 8 years old.
* Elective non complicated adenotonsillectomy.
* ASA I or II physical status.

Exclusion Criteria:

* Refusal of the patient's parents or legal guardians to give informed consent.
* History of allergy to any of the study drugs.
* Preoperative intake of opioid or non-steroidal anti-inflammatory drugs within 24 h before surgery.
* Neurological and/or psychological diseases.
* Associated cardio-respiratory illness

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 222 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
measure sedative effectes of Dexmedetomidine, Ketamine, or Midazolam using modified observer's assessment of alertness/sedation scale and parental separation anxiety scale. | 12 months
  measure sedative effectes of Dexmedetomidine, Ketamine, or Midazolam using modified observer's assessment of alertness/sedation scale and parental separation anxiety scale.

SECONDARY OUTCOMES:
Amount of analgesia required postperative by Face, Legs, Activity, Cry, Consolability (FLACC) Behavioural Pain Scale. | 12 months
  Amount of analgesia required postperative (Analgesia is maintained using diclofenac 1 mg/kg suppository. If 7-10 severe discomfort pain in the FLACC behavioral pain scale is heard, pethidine 1mg/kg/dose once, will be administered for persistent score in the 12-hour postoperative period.) according to Face, Legs, Activity, Cry, Consolability (FLACC) Behavioural Pain Scale
Measure Emergence agitation by Richmond Agitation-Sedation Scale (RASS) | 12 months
  Measure Emergence agitation during recovery using Emergence agitation and recovery profile will be evaluated using the Richmond Agitation-Sedation Scale (RASS) to evaluate the patients' recovery profile.

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia university hospitails, Shibīn al Kawm, Menoufia, Egypt